CLINICAL TRIAL: NCT03174132
Title: A Randomised, Multi-center, Subject and Evaluator-blinded Study Comparing the Pain and the Safety Profile Associate With Correction of Moderate to Severe Nasolabial Folds Using Restylane Perlane Lidocaine Compared to Restylane Perlane
Brief Title: Pain and Safety of Restylane Perlane With and Without Lidocaine for Correction of Moderate and Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43TW1628
Record Dates: First submitted 2017-05-29; First posted 2017-06-02 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-08

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Perlane Lidocaine (Experimental): Restylane Perlane Lidocaine will be injected into one side of the nasolabial fold at day 1
  Interventions: Device: Restylane Perlane Lidocaine
- Restylane Perlane (Active Comparator): Restylane Perlane will be injected into the opposite side of the nasolabial fold on day 1
  Interventions: Device: Restylane Perlane

INTERVENTIONS:
Device: Restylane Perlane Lidocaine — Intradermal injection
  Arms: Restylane Perlane Lidocaine
Device: Restylane Perlane — Intradermal injection
  Arms: Restylane Perlane

SUMMARY:
The purpose of this study is to evaluate the pain and safety in associated with injection of Restylane Perlane Lidocaine compared to Restylane Perlane using VAS scale

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent to participate in the study.
* Men or women aged 20 years or older of Chinese origin.
* Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study.
* Intent to undergo correction of both nasolabial folds (NLF) with a wrinkle severity in Wrinkle Severity Rating Scale (WSRS) of either grade 3 on both NLFs or grade 4 on both NLFs.

Exclusion Criteria:

* Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the lower orbital rim.
* Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim within 12 months before treatment.
* Previous tissue revitalization treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling or dermabrasion in the midface within 6 months before treatment.
* Scars or deformities, active skin disease, inflammation or related conditions near or in the area to be treated.
* Other condition preventing the subject from entering the study in the Investigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University, Kaohsiung City
  - Chang Gung Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane Perlane Lidocaine and Restylane Perlane: Restylane Perlane Lidocaine will be injected into one side of the nasolabial fold at day 1
  Restylane Perlane Lidocaine: Intradermal injection
  Restylane Perlane will be injected into the opposite side of the nasolabial fold on day 1
  Restylane Perlane: Intradermal injection
Period: Overall Study
Arm/Group | Restylane Perlane Lidocaine and Restylane Perlane
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restylane Perlane Lidocaine and Restylane Perlane
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 70
Region of Enrollment [Number; unit: participants]
  Taiwan | 70

OUTCOME MEASURES:

1. Primary Outcome: Treatment Differences in Pain (Restylane Perlane Side - Restylane Perlane Lidocaine Side) as Measured by a Visual Analogue Scale (VAS)
Description: Subjects that reported at least 10 mm less VAS pain associated with injections of Perlane-Lido compared to Perlane at the time of injection.
  VAS=Visual Analogue Scale. The VAS is a subjective scale to measure pain intensity. The participant is instructed to put a vertical mark, approximating the pain experienced during the procedure, on a 100 mm (millimeter) horizontal line labelled "no pain" at the left end and "the worst pain you can imagine" at the right end. The distance in mm from the left end (no pain) to the participant's VAS mark is measured with a standard ruler.
Time Frame: At the time of injection
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Restylane Perlane Lidocaine and Restylane Perlane
Number analyzed (Participants) | 70
percentage of subjects | 87.1 [77.0 to 93.9]

2. Secondary Outcome: Treatment Differences in Pain (Restylane Perlane Side - Restylane Perlane Lidocaine Side) as Measured by a Visual Analogue Scale (VAS)
Description: Subjects that reported at least 10 mm less VAS pain associated with injections of Perlane-Lido compared to Perlane at 15, 30, 45 and 60 minutes after injection.
  VAS=Visual Analogue Scale. The VAS is a subjective scale to measure pain intensity. The participant is instructed to put a vertical mark, approximating the pain experienced during the procedure, on a 100 mm (millimeter) horizontal line labelled "no pain" at the left end and "the worst pain you can imagine" at the right end. The distance in mm from the left end (no pain) to the participant's VAS mark is measured with a standard ruler.
Time Frame: 15, 30, 45, and 60 minutes after injection
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Restylane Perlane Lidocaine and Restylane Perlane
Number analyzed (Participants) | 70
percentage of subjects
  after 15 minutes | 64.3 [51.9 to 75.4]
  after 30 minutes | 42.9 [31.1 to 55.3]
  after 45 minutes | 31.4 [20.9 to 43.6]
  after 60 minutes | 24.3 [14.8 to 36]

ADVERSE EVENTS:
Time Frame: Maximum 32 days for each participant (from screening visit to last visit).
Description: AEs collection began after the informed consent form had been signed. Each subject was questioned about AEs at each clinical visit following the screening visit. The question asked was "Since your last clinical visit have you had any health problems?" Information on AEs could also be obtained from signs and symptoms detected during each examination or from a laboratory test, observations by the study personnel, subject diaries or spontaneous reports from the subjects.
Arm/Group | Restylane Perlane Lidocaine and Restylane Perlane
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 7/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Perlane Lidocaine and Restylane Perlane (N=70)
Presyncope (Nervous system disorders) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT03174132/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03174132/SAP_001.pdf